CLINICAL TRIAL: NCT05115799
Title: Effects of a Manual Therapy Program to Reduce the Evolution Time of Axillary Web Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Jesús Baltasar, Principal Investigator, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AWS
Record Dates: First submitted 2021-10-06; First posted 2021-11-10 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Mastectomy; Lymphedema; Thrombi; Thrombosis; Shoulder Syndrome; Movement Disorders
Keywords: mastectomy; breast cancer; lymphedema; kinesiology applied; thrombosis; health education; rehabilitation
MeSH Terms: conditions — Breast Neoplasms; Lymphedema; Thrombosis; Movement Disorders; Health Education | interventions — Musculoskeletal Manipulations; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Investigator
Masking Description: The randomization of the sample is done through the Excel program, where the "randomization" function distributes the numbers from 1 to 46 (number of research members) in the control group or intervention group.
  As patients with this health problem arrive, they are distributed in order of arrival in both groups as determined by randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Axilliary Web Syndrome and manual therapy and scar massage. (Experimental): These users will come from the first moment of the diagnosis of the thrombus in our unit, to receive manual therapy by the physical therapist. They will receive 15 sessions of manual therapy by the physiotherapist, 5 days a week, each session being approximately 40 minutes long. The session will begin with pendulum exercises of the shoulder to warm up the joint and give proprioceptive stimulation to the joint capsule. The physiotherapist will perform passive stretches looking to put tension on the cord lymphatic, never exceeding grade 6 VAS pain. Mainly the shoulder will be worked affected, and if the cord reaches the crease of the elbow or thumb, the extension-supination of the elbow, and ulnar deviation of the wrist.
  Scar massage will be done in the area where the lymphatic cord originates at the proximal level while maintaining the tolerable tension of the lymphatic cord (during the massage also pain grade 6 VAS will be exceeded).
  Interventions: Other: Manual Therapy, Physiotherapy, Kinesiology, Scar Massage
- Patients with Axilliary Web Syndrome and health education and kinesiotherapy. (Other): These users will be instructed in hygienic-postural care and active auto-kinesitherapy assisted to perform daily for 30 minutes. The investigators will value following the instructions every 30 days
  Interventions: Other: Kinesiotherapy, Physiotherapy, Health Education

INTERVENTIONS:
Other: Manual Therapy, Physiotherapy, Kinesiology, Scar Massage — The physiotherapist performs passive kinesitherapy on the mastectomized patient with lymphatic thrombus, and scar massage when the arm maintains its greater range of mobility.
  The patient will never present pain during the rehabilitation session above 5 in Pain Scale Analog Scale.
  Arms: Patients with Axilliary Web Syndrome and manual therapy and scar massage.
Other: Kinesiotherapy, Physiotherapy, Health Education — These users will be instructed in hygienic-postural care and active auto-kinesitherapy assisted to perform daily for 30 minutes. The investigators will value following the instructions every 30 days
  Arms: Patients with Axilliary Web Syndrome and health education and kinesiotherapy.

SUMMARY:
ABSTRACT

Breast cancer is the most common malignant tumor in women, with more than a million new cases annually. One of the most frequent surgical and post-actinic sequelae and well known is postmastectomy lymphedema. The axillary web syndrome is another sequel that limits the functionality of the patient and delays the protocol times of application of treatments cancer, and in many cases this sequela is misdiagnosed. This surgical sequelusually disappears spontaneously after the third month of appearance, but this implies a long period of discomfort and limitations for the user, at the same time that it may delay the application of Radiotherapy within the indicated protocol deadlines (due to the need for a body posture with abduction and flexion of the affected upper limb for its application and with the lymphatic thrombus is impossible to get).

With the present quasi-experimental study, the investigator intend to show that the application of Kinesitherapy and stretching from the beginning of the appearance of the cord, in a controlled and scheduled way by the physiotherapist, it is possible to reduce the time in which the lymphatic thrombus is present, and therefore, recover functionality, mobility, reduce pain and be able to apply the patients´ treatments within of the established deadlines. The investigator intend to apply this therapy in the intervention group and compare thrombus evolution times with the control group.

DETAILED DESCRIPTION:
BACKGROUND AND CURRENT STATUS OF THE STUDY TOPIC

Breast Cancer is the most common tumor in women around the world, and is one of the leading causes of death among women in developed countries.

It is an important Public Health problem, since according to the World Health Organization more than a million new cases are diagnosed annually, becoming almost a quarter of malignant tumors in females. In the West, it has been shown that one in nine to twelve women will suffer from the disease in her lifetime.

Most cases occur in postmenopausal women, and the main age at diagnosis is around 60 years.

After the diagnosis of breast cancer, the patient undergoes surgical and / or cancer treatment. Chemotherapy, radiotherapy and hormonal therapy are some of the treatment alternatives, which currently are precisely adapted to the type of tumor seeking a better response and survival.

Postmastectomy lymphedema is one of the best-known postsurgical and post-actinic sequelae after breast cancer, with a prevalence of around 20% of mastectomized women.

The conservative treatment of this health problem is based on Decongestive Physical Therapy and Kinesitherapy. Pneumatic Multicompartmental Pressotherapy helps reduce the feeling of heaviness and stiffness of edema.

In addition to postmastectomy lymphedema, the patient undergoing surgery for breast cancer may present Axillary Web Syndrome (AWS) or superficial lymphatic thrombosis. As described by W.M. Yeung et al. In their systematic review, it can appear in the first eight weeks after the operation and usually resolves spontaneously within three months of its appearance.

The lymphatic thrombus is clinically manifested as a cord that frequently occurs in the armpit, although it can also appear along the upper limb, elbow crease even reaching the first finger. Regarding the diagnosis through imaging tests, nuclear magnetic resonance does not manage to clearly identify the axillary network syndrome, being ultrasound the most reliable method, due to the dynamism that can be applied to the patient's arm while the diagnostic test is being carried out.

The axillary network syndrome produces pain when abducting and flexing the shoulder, with the respective loss of functionality and limitation of mobility of the affected upper limb.

According to the American Cancer Society, radiation therapy is applied 3-8 weeks after the operation if chemotherapy is not required. If chemotherapy is used, it is applied 3-4 weeks after completion. It is usually applied 5 days a week from Monday to Friday.

The limitation of mobility often leads to a delay in the application of this useful tool in the oncological therapeutic arsenal to prevent recurrences. Hence, the need and importance of this study, where the investigator intend to demonstrate that the evolution times of the lymphatic thrombus can be reduced with assisted passive kinesitherapy and stretching.

At present, there are some publications that show possible alternatives of physiotherapy treatment for lymphatic thromb. Many are interventions with a very small sample (even on a caseby-case basis). Others are observational studies or even studies older than five years. There are some studies that combine manual lymphatic drainage (Vodder method) with physical therapy (strengthening, stretching, soft tissue work) with good results.

There is ambiguity in the relationship-association between the appearance of lymphatic thrombosis and lymphedema of the ipsilateral limb. Patients who have developed AWS are 44% more likely to develop postmastectomy lymphedema. There are other studies that do not find a relationship between the two.

The frequency of the AWS is not clear from the current posts. It depends on the type of surgical intervention, age, BMI, the appearance of the postoperative seroma, and even breast reconstruction. Thus being the frequency 30% of the operated patients.

After reviewing the relevant literature, it should be noted that there are very few studies and therefore little evidence on the treatment of AWS. It is not possible to prescript of a clear treatment in a clinical practice guide for this postsurgical sequela. Most publications highlight the importance and need for more research to determine the etiopathogenesis and useful treatment for this health issue.

OBJECTIVES GENERAL OBJECTIVES

I. Determine a preliminary exploration of the magnitude of the effect of a kinesitherapy and stretching intervention for the functional recovery of the upper limb, the recovery of the surgical scar and the improvement of the quality of life in women who have suffered from breast cancer. II. Create a scale to objectively classify the axillary thrombus (based on its clinical manifestations).

SPECIFIC OBJECTIVES for general objective I:

* Check the intervention of assisted passive kinesitherapy and stretching for the improvement of the range of joint mobility of the affected limb in the shortest possible time. - Analyze the reduction of pain and increase of the degree of functionality of the ipsilateral upper limb in patients with AWS after the intervention.
* Determine the impact of the physiotherapeutic intervention on the quality of life of a mastectomized woman with lymphatic thrombus.
* Analyse the physiotherapeutic intervention reduction of the time on the evolution of the Superficial Lymphatic Thrombus and the application of Radiotherapy within the terms established in the oncological protocols.

SPECIFIC OBJECTIVES for general objective II:

- Create a scale to objectively classify the axillary thrombus (based on its clinical manifestations).

METHODOLOGY TYPE OF STUDY

Quasi-experimental, prospective study.

STUDY POPULATION

The study sample is made up of patients undergoing surgery for Breast Cancer who attend the Lymphedema Unit of the A.G.S. Campo de Gibraltar Oeste presenting Lymphatic Thrombus after the operation, the recruitment period being from December 2021 to December 2023.

DESCRIPTION OF THE INTERVENTION

15 sessions of Assisted Passive Kinesitherapy are carried out by the physiotherapist. Five days a week, for three weeks. If it is previously referred, the treatment will be finished earlier (the patient must achieve the same ranges of motion and strength as the contralateral limb, together with the remission of pain).

The stretches applied during the sessions will be gentle and maintained, never exceeding a pain grade 5 VAS (moderate pain), once the tension of the cord is reached between 20-30 seconds. A special effort will be made to recover flexion and abduction of the shoulder, bringing the cord to a tolerable tension on the part of the patient.

Friction will be made on the axillary scar to dislodge underlying planes and the subcutaneous tissue of the muscle fascia.

The patient will be trained in active kinesitherapy to prevent lymphedema and activate lymphatic circulation. Also with hygienic-postural measures for the same purpose.

CONTROL GROUP

All the variables and data for each patients are recorded in their clinical history. Goniometric study will be performed of the affected upper limb (shoulder, elbow, wrist). Constant scale, Quick-Dash, the Visual Analog Pain Scale and the International Scale of Physical Activity will also be performed. This assessment will be carried out the patient arrives at our unit and on day 30, 60, 90.

These patients will be instructed in hygienic-postural care and active assisted autokinesitherapy to perform daily for 30 minutes. It will be assessed every 30 days.

These exercises are explained to the patient to be executed at home.

INTERVENTION GROUP

As well as the control group, all the variables and data for each patient will be collected in their medical history. Goniometric study of the affected upper limb will be performed too (shouderelbow-wrist). Constan scale, Quick- DASH, Visual Scale will also be completed together with Analogue of Pain and the International Scale of Physical Activity. This exploration will also take place during the first session and on the 30th, 60th and 90th day.

These users will arrive at the first diagnosis of the thrombus in our unit,in order to receive manual therapy by the physical therapist. (see therapy pictures).

They will receive 15 sessions of manual therapy the physiotherapist, 5 days a week ,each session being approximately 40 minutes long.

The session will begin with pendulum exercises of the shoulder to warm up the joint and give proprioceptive stimulation to the joint capsule.

The physiotherapist will perform passive stretches looking to tensioning the lymphatic cord, never exceeding grade 6 VAS pain chart. Mainly the affected shoulder will be treated and if the cord reaches the crease of the elbow or thumb, the extension (frase sin sentido general hay que volverla a escribir).

Scar massage will be done in the area where the lymphatic cord originates at the proximal level while maintaining the tolerable tension of the lymphatic cord (during the massage also pain grade 6VAS will be exceeded).

Patients with developed lymphedema will receive Decongestive Physical Therapy (PDT) on the treated limb once the 15 day treatment described for the study is finished. Therefore, PDT does not influence on obtained contaminated results. Those patients who do not suffer from lymphedema do not receive PDT.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old.
* Mastectomized patients (either radical or conservative surgery).
* Patient with lymphatic thrombus in the upper limb ipsilateral to the surgical intervention.

Exclusion Criteria:

* Significant psychological alterations that would prevent the retrieval of the information necessary for the investigation.
* Significant neurological alterations that would prevent the retrieval of the information necessary for the investigation.
* Patients in a situation of legal dispute that would affect their intervention in this study.
* Metastasis not treated with chemotherapy treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-04 (Estimated)

PRIMARY OUTCOMES:
Shoulder Range of Movement (ROM) in the limb with Axillary Web Syndrome | 3 Months
  The investigators will use Goniometry of both shoulders. It is a continuous quantitative variable. Goniometer is the standard instrument for measuring the range of movement. The patients were asked to move thir arms in flexion, extension, abduction and external and internal rotation of the shoulder. It was considered that the maximum range of motion for the flexion and abduction was 180º, for extension it was 45º, 100º for internal rotation and 80º for external rotation. Finally, a single index was calculated as the percentage of global movement ().
Quality of life. Barthel Scale | 3 Months
  The investigators will use the Barthel Scale.
  The Barthel index or Barthel scale is an instrument used by social and health professionals for the functional assessment of a patient and to monitor their evolution. In the case of Social Workers, they value the independence or dependence of the person in each of the activities of daily living (ADL), obtaining as a result the level of performance of the person and carrying out a rehabilitative / compensatory intervention and / or maintenance according to the results obtained. Promoting and / or maintaining the independence of the person.
  The scale measures the ability of a person to perform 10 activities of daily life, which are considered basic, in this way a quantitative estimate of their degree of independence is obtained. 100 points is the highest score and the best result in the patient's functionality. 0 points is the worst result and shows the worst functional status.

SECONDARY OUTCOMES:
Shoulder Functionality tested with DASH Scale | 3 Months
  The investigators will use the DASH Scale.
  The Disabilities of the Hand, Arm and Shoulder (DASH) questionnaire is a specific instrument for measuring the quality of life related to health problems to the upper limbs. It is validated in Spanish and it consists of 30 questions. The final score calculation is relatively complicated. In order to calculate the scores it is necessary to have answered at least 27 out of the 30 questions. The final scores is obtained by calculating the arithmetic means of the questions answered minus 1 times 25. The DASH questionnaire has excellent reproductibility and high sensitivity, being able to detect small changes. The scale ranges from 30 to 150 points. 30 points means good shoulder functionality and 150 non-functional shoulder.
  It has two optional subsections where sports and work functionality can be assessed.
Shoulder Pain. Visual Analogic Scale (VAS) | 3 Months
  The investigators will use the Visual Analog Pain Scale.
  According to the National Cancer Institue ( NIH), it is a tool used to help the professional assess the intensity of certain sensations and feelings, such as pain. The Visual Analog Scale for pain is composed of a straight line on which an extreme means no pain and the other extreme means the worst pain imaginable.
  Extreme pain corresponds to 10 points. None pain corresponds to 0 points.
  The patient marks a point on the line that matches the amount of pain they feel. Also known as VAS.
Shoulder Functionality tested with Constant Scale | 3 Months
  The investigators wil use the Constant Scale. Constant Scale: According to the Spanish Society for Shoulder and Elbow Surgery (SECHC), the Constant Scale assesses pain, functionality for daily life activities, joint mobility and shoulder strength. Also, it considers the laterality and the time it takes the patient. The score ranges from 0 points to 100 points, being 100 the optimal condition for the shoulder.

CONTACTS AND LOCATIONS:
Overall Officials: Rocío Martín Valero, Physiothera, Study Director — Malaga U; María Jesús Viñolo Gil, Physiothera, Study Director — Cádiz U
Locations (1):
- Jesús Baltasar González Rubiño, Algeciras, Cádiz, Spain

IPD SHARING:
Plan to Share IPD: Yes
1. Publication in journals indexed in the Journal Citation Report (JCR), in the field of Oncology and Rehabilitation and Physical Medicine and Physiotherapy.
  2. Dissemination of results in national and international Congresses of Oncology and Rehabilitation and Physical Medicine and Physiotherapy.
  3. Dissemination to the public, press releases and explanatory brochures of the project.
  4. Dissemination on the website of the A.G.S. Campo de Gibraltar West.
Supporting Information: ICF, CSR
Time Frame: In two years. In October 2023.
Access Criteria: Open file

REFERENCES:
- [Result] Sancho-Garnier H, Colonna M. [Breast cancer epidemiology]. Presse Med. 2019 Oct;48(10):1076-1084. doi: 10.1016/j.lpm.2019.09.022. Epub 2019 Nov 6. French. PMID 31706896
- [Result] Waks AG, Winer EP. Breast Cancer Treatment: A Review. JAMA. 2019 Jan 22;321(3):288-300. doi: 10.1001/jama.2018.19323. PMID 30667505
- [Result] Gillespie TC, Sayegh HE, Brunelle CL, Daniell KM, Taghian AG. Breast cancer-related lymphedema: risk factors, precautionary measures, and treatments. Gland Surg. 2018 Aug;7(4):379-403. doi: 10.21037/gs.2017.11.04. PMID 30175055
- [Result] Shao Y, Zhong DS. Manual lymphatic drainage for breast cancer-related lymphoedema. Eur J Cancer Care (Engl). 2017 Sep;26(5). doi: 10.1111/ecc.12517. Epub 2016 May 11. PMID 27167238
- [Result] Soriano-Maldonado A, Carrera-Ruiz A, Diez-Fernandez DM, Esteban-Simon A, Maldonado-Quesada M, Moreno-Poza N, Garcia-Martinez MDM, Alcaraz-Garcia C, Vazquez-Sousa R, Moreno-Martos H, Toro-de-Federico A, Hachem-Salas N, Artes-Rodriguez E, Rodriguez-Perez MA, Casimiro-Andujar AJ. Effects of a 12-week resistance and aerobic exercise program on muscular strength and quality of life in breast cancer survivors: Study protocol for the EFICAN randomized controlled trial. Medicine (Baltimore). 2019 Nov;98(44):e17625. doi: 10.1097/MD.0000000000017625. PMID 31689771
- [Result] Tastaban E, Soyder A, Aydin E, Sendur OF, Turan Y, Ture M, Bilgen M. Role of intermittent pneumatic compression in the treatment of breast cancer-related lymphoedema: a randomized controlled trial. Clin Rehabil. 2020 Feb;34(2):220-228. doi: 10.1177/0269215519888792. Epub 2019 Dec 4. PMID 31795748
- [Result] Yeung WM, McPhail SM, Kuys SS. A systematic review of axillary web syndrome (AWS). J Cancer Surviv. 2015 Dec;9(4):576-98. doi: 10.1007/s11764-015-0435-1. Epub 2015 Feb 15. PMID 25682072
- [Result] Furlan C, Matheus CN, Jales RM, Derchain S, Sarian LO. Vascular Alterations in Axillary and Brachial Vessels in Patients with Axillary Web Syndrome After Breast Cancer Surgery. Lymphat Res Biol. 2018 Jun;16(3):287-293. doi: 10.1089/lrb.2017.0037. Epub 2017 Sep 29. PMID 28961070
- [Result] Leduc O, Fumiere E, Banse S, Vandervorst C, Clement A, Parijs T, Wilputte F, Maquerlot F, Ezquer Echandia M, Tinlot A, Leduc A. Identification and description of the axillary web syndrome (AWS) by clinical signs, MRI and US imaging. Lymphology. 2014 Dec;47(4):164-76. PMID 25915977
- [Result] Jacob T, Bracha J. Identification of Signs and Symptoms of Axillary Web Syndrome and Breast Seroma During a Course of Physical Therapy 7 Months After Lumpectomy: A Case Report. Phys Ther. 2019 Feb 1;99(2):229-239. doi: 10.1093/ptj/pzy110. PMID 30339213
- [Result] Koehler LA, Hunter DW, Haddad TC, Blaes AH, Hirsch AT, Ludewig PM. Characterizing axillary web syndrome: ultrasonographic efficacy. Lymphology. 2014 Dec;47(4):156-63. PMID 25915976
- [Result] Baggi F, Nevola Teixeira LF, Gandini S, Simoncini MC, Bonacossa E, Sandrin F, Sciotto Marotta M, Lanni G, Dadda P, Colpani D, Luini A. Axillary web syndrome assessment using a self-assessment questionnaire: a prospective cohort study. Support Care Cancer. 2018 Aug;26(8):2801-2807. doi: 10.1007/s00520-018-4123-3. Epub 2018 Mar 5. PMID 29508139
- [Result] Huang HC, Liu HH, Yin LY, Weng CH, Fang CL, Yang CS. High Incidence of Axillary Web Syndrome among Breast Cancer Survivors after Breast Reconstruction. Breast Care (Basel). 2020 Aug;15(4):366-371. doi: 10.1159/000501928. Epub 2019 Nov 12. PMID 32982646
- [Result] Ramirez-Parada K, Garay-Acevedo D, Mella-Abarca W, Petric-Guajardo M, Sanchez-Rojel C, McNeely ML, Leao-Ribeiro I, Fernandez-Verdejo R. Axillary web syndrome among Chilean women with breast cancer: incidence and possible predisposing factors. Support Care Cancer. 2020 Jun;28(6):2941-2947. doi: 10.1007/s00520-019-05190-5. Epub 2019 Nov 25. PMID 31768730
- [Result] Koehler LA, Blaes AH, Haddad TC, Hunter DW, Hirsch AT, Ludewig PM. Movement, Function, Pain, and Postoperative Edema in Axillary Web Syndrome. Phys Ther. 2015 Oct;95(10):1345-53. doi: 10.2522/ptj.20140377. Epub 2015 May 14. PMID 25977305
- [Result] Yao Y, Chu Y, Xu B, Hu Q, Song Q. Radiotherapy after surgery has significant survival benefits for patients with triple-negative breast cancer. Cancer Med. 2019 Feb;8(2):554-563. doi: 10.1002/cam4.1954. Epub 2019 Jan 10. PMID 30632300
- [Result] Hickey BE, Francis DP, Lehman M. Sequencing of chemotherapy and radiotherapy for early breast cancer. Cochrane Database Syst Rev. 2013 Apr 30;(4):CD005212. doi: 10.1002/14651858.CD005212.pub3. PMID 23633328
- [Result] White JR, Meyer JL. Intensity-modulated radiotherapy for breast cancer: advances in whole and partial breast treatment. Front Radiat Ther Oncol. 2011;43:292-314. doi: 10.1159/000322461. Epub 2011 May 20. PMID 21625159
- [Result] Xu HP, Bronsart E, Costa E, Krhili S, Logerot C, Bazire L, Fournier-Bidoz N, Belshi A, Fourquet A, Kirova YM. Patterns of locoregional failure in women with early-stage breast cancer treated by whole breast irradiation in the lateral isocentric decubitus position: Large-scale single-centre experience. Cancer Radiother. 2019 Apr;23(2):116-124. doi: 10.1016/j.canrad.2018.08.002. Epub 2019 Mar 29. PMID 30935887
- [Result] Fourie WJ, Robb KA. Physiotherapy management of axillary web syndrome following breast cancer treatment: discussing the use of soft tissue techniques. Physiotherapy. 2009 Dec;95(4):314-20. doi: 10.1016/j.physio.2009.05.001. Epub 2009 Jul 29. PMID 19892098
- [Result] Cho Y, Do J, Jung S, Kwon O, Jeon JY. Effects of a physical therapy program combined with manual lymphatic drainage on shoulder function, quality of life, lymphedema incidence, and pain in breast cancer patients with axillary web syndrome following axillary dissection. Support Care Cancer. 2016 May;24(5):2047-2057. doi: 10.1007/s00520-015-3005-1. Epub 2015 Nov 5. PMID 26542271
- [Result] Ryans K, Davies CC, Gaw G, Lambe C, Henninge M, VanHoose L. Incidence and predictors of axillary web syndrome and its association with lymphedema in women following breast cancer treatment: a retrospective study. Support Care Cancer. 2020 Dec;28(12):5881-5888. doi: 10.1007/s00520-020-05424-x. Epub 2020 Apr 8. PMID 32270312
- [Result] Wariss BR, Costa RM, Pereira AC, Koifman RJ, Bergmann A. Axillary web syndrome is not a risk factor for lymphoedema after 10 years of follow-up. Support Care Cancer. 2017 Feb;25(2):465-470. doi: 10.1007/s00520-016-3424-7. Epub 2016 Oct 4. PMID 27704260
- [Result] Fisher MI, Capilouto G, Malone T, Bush H, Uhl TL. Comparison of Upper Extremity Function in Women With and Women Without a History of Breast Cancer. Phys Ther. 2020 Mar 10;100(3):500-508. doi: 10.1093/ptj/pzaa015. PMID 32031629
- [Result] Celik D, Kaya Mutlu E. Does adding mobilization to stretching improve outcomes for people with frozen shoulder? A randomized controlled clinical trial. Clin Rehabil. 2016 Aug;30(8):786-94. doi: 10.1177/0269215515597294. Epub 2015 Jul 30. PMID 26229109
- [Result] Budtz CR, Andersen JH, de Vos Andersen NB, Christiansen DH. Responsiveness and minimal important change for the quick-DASH in patients with shoulder disorders. Health Qual Life Outcomes. 2018 Dec 10;16(1):226. doi: 10.1186/s12955-018-1052-2. PMID 30526622
- [Result] Vrotsou K, Avila M, Machon M, Mateo-Abad M, Pardo Y, Garin O, Zaror C, Gonzalez N, Escobar A, Cuellar R. Constant-Murley Score: systematic review and standardized evaluation in different shoulder pathologies. Qual Life Res. 2018 Sep;27(9):2217-2226. doi: 10.1007/s11136-018-1875-7. Epub 2018 May 10. PMID 29748823
- [Result] Hervas MT, Navarro Collado MJ, Peiro S, Rodrigo Perez JL, Lopez Mateu P, Martinez Tello I. [Spanish version of the DASH questionnaire. Cross-cultural adaptation, reliability, validity and responsiveness]. Med Clin (Barc). 2006 Sep 30;127(12):441-7. doi: 10.1157/13093053. Spanish. PMID 17040628
- [Result] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588
- [Result] Arraras JI, Asin G, Illarramendi JJ, Manterola A, Salgado E, Dominguez MA. The EORTC QLQ-ELD14 questionnaire for elderly cancer patients. Validation study for elderly Spanish breast cancer patients. Rev Esp Geriatr Gerontol. 2019 Nov-Dec;54(6):321-328. doi: 10.1016/j.regg.2019.05.001. Epub 2019 Jun 30. PMID 31266659
- [Derived] Gonzalez-Rubino JB, Martin-Valero R, Vinolo-Gil MJ. Physiotherapy protocol to reduce the evolution time of axillary web syndrome in women post-breast cancer surgery: a randomized clinical trial. Support Care Cancer. 2025 Mar 28;33(4):326. doi: 10.1007/s00520-025-09373-1. PMID 40153020
- [Derived] Gonzalez Rubino JB, Vinolo-Gil MJ, Garcia Munoz C, Martin-Valero R. Randomised clinical trial of a manual therapy programme to reduce the evolution time of axillary web syndrome in women affected by breast cancer: study protocol. BMJ Open. 2022 Sep 21;12(9):e063305. doi: 10.1136/bmjopen-2022-063305. PMID 36130744
- See also: Pain Visual Analogic Score — https://www.cancer.gov/espanol/publicaciones/diccionarios/diccionario-cancer/def/escala-visual-analogica
- See also: Constant Score Test for Shoulder — https://sechc.es/test-score-hombro/603-constant-score-test-valoracion-hombro
- See also: Calculation of the sample size — https://www.fisterra.com/formacion/metodologia-investigacion/determinacion-tamano-muestral/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/99/NCT05115799/Prot_SAP_ICF_000.pdf